CLINICAL TRIAL: NCT06338527
Title: Effects of Aromatherapy on Sleep Quality and Anxiety in Patients Undergoing Chemotherapy for Breast Cancer
Brief Title: Effects of Aromatherapy on Patients Undergoing Chemotherapy for Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weifang Medical University (Other)
Responsible Party: Principal Investigator, Jiang Liu, Research investigator, Weifang Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024YX321
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Sleep Quality; Anxiety
Keywords: Sleep quality; Anxiety; Aromatherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): The researchers placed 2 drops of lavender oil on gauze in a box each night 30 minutes before the patient went to bed and placed it 15 to 20 centimeters from the pillow.
  Interventions: Other: Aromatherapy
- Control group (Active Comparator): The control group had no aromatherapy intervention during the study period.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Aromatherapy — Lavender oil was used for aromatherapy intervention.
  Arms: Experimental group
Other: No intervention — No aromatherapy intervention was performed during the period of the study.
  Arms: Control group

SUMMARY:
The objective of this study was to investigate the effects of aromatherapy on sleep quality and anxiety in patients undergoing chemotherapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria: 1) patients diagnosed with breast cancer and receiving chemotherapy; 2) suffering from sleep disorders or PSQI score greater than 5; 3) not using medications such as antidepressants and hypnotics that may affect the observation results; 4) age older than 18 years and volunteered to participate in this study.

Exclusion Criteria: 1) Asthma or severe respiratory disease; 2) Allergy to lavender; 3) Cognitive or communication disorders; 4) Breast cancer combined with severe organ dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-26 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | The sleep quality of the patients was assessed at 8 a.m. for one week.
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess the sleeping quality of the patients. The total score of PSQI ranged from 0-21, with higher scores indicating poor sleep quality.
Anxiety | The anxiety level of the patients was assessed at 8 a.m. for one week.
  Beck Anxiety Inventory (BAI) was used to assess the anxiety level of the patients. The scale consists of 21 entries with a total score ranging from 0 to 63, with higher total scores being associated with more severe levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Shirong Fang, M.D., Principal Investigator — Weifang People's Hospital
Locations (1):
- Weifang People's Hospital, Weifang, Shangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang F, Cheng L, Qin S, Wang L, Liu Y, Liu Y, Yang J, Fang S, An N, Zhang Y, Liu J. Effect of aromatherapy massage with lavender essential oil on sleep quality, pain, and mental and psychiatric disorders among breast cancer patients undergoing chemotherapy: a randomized controlled trial. Support Care Cancer. 2025 Jul 14;33(8):689. doi: 10.1007/s00520-025-09741-x. PMID 40653563